CLINICAL TRIAL: NCT03419598
Title: Personalised Subject Specific HTO Versus Generic HTO Virtual Clinical Trial
Brief Title: Personalised HTO Versus Generic HTO Virtual Clinical Trial
Status: Completed | Type: Observational
Sponsor: University of Bath (Other)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Richie Gill, Professor, University of Bath
Other Study IDs: RG433_TVT003
Record Dates: First submitted 2018-01-26; First posted 2018-02-05 (Actual); Results first posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis, Knee
Keywords: virtual clinical trial; high tibial osteotomy; 3D; computer simulation; finite element analysis; medial unicompartmental knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All study participants: All virtual participants who received a virtual opening wedge high tibial osteotomy. The baseline information was the individual CT-based geometry of tibia.
  Interventions: Procedure: Opening wedge high tibial osteotomy; Device: Personalised subject specific custom HTO plate; Device: Generic HTO plate

INTERVENTIONS:
Procedure: Opening wedge high tibial osteotomy — Realignment of knee by creating an opening wedge osteotomy in the upper part of the tibia. Since this is a virtual trial, the virtual patients were duplicated and enrolled into both arms
  Other Names: HTO
Device: Personalised subject specific custom HTO plate — Subject specific custom plate for stabilizing an open wedge HTO
  Other Names: Personalised plate
Device: Generic HTO plate — Generic plate for stabilizing an open wedge HTO
  Other Names: Generic plate

SUMMARY:
High Tibial Osteotomy (HTO) is an alternative to knee replacement in suitable patients with early knee osteoarthritis (OA), it is particularly suited to patients with single compart disease who otherwise would be suitable for unicompartmental knee replacement (UKR). OA of the knee is very common and increasing driven by the ageing of the population. The current limitations of HTO are related to the difficulty of achieving the desired correction due to a challenging surgical technique and soft tissue irritation due to the use of generic stabilisation plates. This study will examine the safety equivalence of a new patient specific HTO process which has patient specific 3D printed plates, i.e. personalised HTO plates, with the existing most commonly used HTO procedure using the Tomofix generic HTO plate. Importantly this study will be undertaken as a Virtual Trial, existing anonymised 3D imaging data will be used to create the virtual patient cohort. This cohort will receive both procedures, which for this type of procedure is only possible in a virtual scenario.

The main question to be addressed is: "Is the personalised HTO procedure as safe as the most commonly used existing generic HTO procedure?". In this context safety concerns the mechanical loads placed upon the tibia and the support plate.

The interventions will all be made on computer models, the 3D imaging data will be used to create the intact (un-operated) models of the subject tibias. Each model will then be virtually operated upon, with both the personalised and generic HTO procedures. The models will then be loaded with physiological loads experienced during function and the mechanical states compared.

DETAILED DESCRIPTION:
Ethical approval was obtained to use CT scans of 30 patients with moderate to severe knee arthritis (REC reference: 17/HRA/0033, Royal Devon & Exeter National Health Service [NHS], UK).

The CT data will be used to generate the 3D geometry of each patient's proximal tibia. The osteotomy correction angle required for each patient such that the altered mechanical axis will pass through a point 62.5% of the distance from medial to lateral tibial plateau. Virtual HTO surgery will be performed on each patient to alter the mechanical axis of the knee by creating an opening wedge osteotomy.

After the virtual surgeries are performed, each virtual patient will be duplicated. One copy will have the osteotomy stabilised using a Generic plate and the other using a Personalised plate, thus forming the two arms of the trial.

For each participant in each arm finite element (FE) models will be created, and loads applied simulating walking, sit to stand and squatting. Four healings stages will be considered, stage 1 being immediately post-operation (this will not be modelled), stage 2 representing 2 weeks post-operation, stage 3 representing 6 weeks and stage 4 representing 12 weeks. The mechanical loads in the plates, and around the screw locations in the bone, will be established by solving these finite element models.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate existing CT data of lower limb.
* Male or Female, aged 18 years or above.
* Diagnosed with moderate to severe OA of the knee.

Exclusion Criteria:

* Abnormal anatomy of tibia or presence of pathology other than OA, e.g. bone tumour.
* Previous knee or osteotomy surgery.
* Presence of metal-work

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population was recruited from waiting list of patients with knee OA
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richie Gill, DPhil, Principal Investigator — University of Bath; Andrew Toms, MD, Principal Investigator — Royal Devon & Exeter NHS Trust
Locations (2):
- United Kingdom (2):
  - Royal Devon & Exeter NHS Trust, Exeter, Devon
  - University of Bath, Bath

IPD SHARING:
Plan to Share IPD: No
Virtual cohort may be re-used for further studies, all virtual patients are anonymized

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The virtual patients were created based on CT data sets obtained for 30 patients with knee osteoarthritis. The virtual patients were duplicated, and then enrolled into both arms.
Groups:
- All Study Participants: Opening wedge high tibial osteotomy (HTO).
  Realignment of knee by creating an opening wedge osteotomy in the upper part of the tibia.
  Since this is a virtual trial, the virtual patients were duplicated and had the osteotomy stabilised by a generic HTO plate in one copy of the cohort and by a personalised HTO plate in the other copy.
Period: Overall Study
Arm/Group | All Study Participants
Started (Since this is a virtual trial, the virtual patients were duplicated and enrolled into both arms) | 30
Subject Specific Tibia Models Created and Virtual Osteotomy Performed | 28
Virtual Cohort Duplicated Into A. Personalised and B. Generic Copies | 28
Finite Element (FE) Model Created for Cohort Copy Stabilised by Personalised HTO Plate | 28
FE Models Created for Cohort Copy Stabilised by Generic HTO Plate | 28
FE Models Solved for Personalised HTO Plate Stabilised Cohort Copy | 28
FE Models Solved for Generic HTO Plate Stabilised Cohort Copy | 28
Completed | 28
Not Completed | 2
Not completed — Poor quality CT scans could not be adequately segmented to create virtual patient tibial geometry | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Opening wedge high tibial osteotomy (HTO): Realignment of knee by creating an opening wedge osteotomy in the upper part of the tibia
  Cohort duplicated into 2 copies. Copy A. Stabilised by Personalised HTO plate. Copy B. Stabilised by Generic HTO plate.
Arm/Group | All Study Participants
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 28
Height (m) [Mean (Standard Deviation); unit: metres] | 1.686 (0.124)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 90.1 (16.4)
Kellgren & Lawrence OA Grade [Mean (Standard Deviation); unit: units on a scale] — Radiographic grading scale for osteoarthritis (OA) of a joint.
  Grade 0 (none): definite absence of x-ray changes of osteoarthritis. Grade 1 (doubtful): doubtful joint space narrowing and possible osteophytic lipping.
  Grade 2 (minimal): definite osteophytes and possible joint space narrowing. Grade 3 (moderate): moderate multiple osteophytes, definite narrowing of joint space and some sclerosis and possible deformity of bone ends.
  Grade 4 (severe): large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends.
  units on a scale | 2.6 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Stress in Plate During Gait
Description: Mechanical stress (Von Mises) calculated for functional loading using finite element analysis
Time Frame: 6 weeks simulated post-operation
Measure: Mean (Standard Error); unit: MPa
Groups:
- Personalised HTO: Opening wedge high tibial osteotomy
  Personalised subject specific custom HTO plate
  Opening wedge high tibial osteotomy: Realignment of knee by creating an opening wedge osteotomy in the upper part of the tibia
  Stabilised by personalised HTO plate, contoured to subject's tibial geometry
- Generic HTO: Opening wedge high tibial osteotomy
  Generic HTO plate
  Opening wedge high tibial osteotomy: Realignment of knee by creating an opening wedge osteotomy in the upper part of the tibia
  Generic HTO plate: Generic plate for stabilizing an open wedge HTO
Arm/Group | Personalised HTO | Generic HTO
Number analyzed (Participants) | 28 | 28
MPa | 108.3 (3.81) | 90.6 (3.56)

2. Secondary Outcome: Mechanical Strain in Bone Around Screws During Gait
Description: Mechanical strain calculated for functional loading using finite element analysis, note strain is dimensionless and hence has no units
Time Frame: 6 weeks simulated post-operation
Measure: Mean (Standard Error); unit: unitless
Groups:
- Personalised HTO: Opening wedge high tibial osteotomy
  Personalised subject specific custom HTO plate
  Opening wedge high tibial osteotomy: Realignment of knee by creating an opening wedge osteotomy in the upper part of the tibia
  Stabilising by personalised HTO contoured to subject's tibial geometry
Arm/Group | Personalised HTO | Generic HTO
Number analyzed (Participants) | 28 | 28
unitless | 0.011 (0.00056) | 0.011 (0.00065)

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed
Description: Adverse Events were not monitored/assessed
Groups:
- All Study Participants: Opening wedge high tibial osteotomy (HTO): Realignment of knee by creating an opening wedge osteotomy in the upper part of the tibia.
  Virtual cohort duplicated into A. stabilised by Personalised HTO plate and B. stabilised by Generic HTO plate.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The main failure mode of HTO plates is fatigue failure, if the peak stress is below the fatigue limit the risk of fatigue failure is low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT03419598/Prot_SAP_000.pdf